CLINICAL TRIAL: NCT02358876
Title: BradyXplore Phase II: Bradykinesia Feature Extraction System
Status: Completed | Type: Observational
Sponsor: Great Lakes NeuroTechnologies Inc. (Industry)
Collaborators: University of Cincinnati (Other); The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 5R44NS065554 (NIH)
Record Dates: First submitted 2015-02-04; First posted 2015-02-09 (Estimated); Results first posted 2016-10-06 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-08

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Deep brain stimulation; Bradykinesia
MeSH Terms: conditions — Parkinson Disease; Hypokinesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Study objectives are to improve motion sensor algorithms for measuring bradykinesia in the clinic and the home, evaluate test-retest reliability of motion sensor algorithms for measuring bradykinesia compared to clinician raters, determine if participant-perceived symptom severities correlate with motion sensor measures, determine if speed, amplitude, and rhythm fluctuate differentially throughout the day in individuals with implanted deep brain stimulation systems, receive feedback on the usability of Kinesia One, and evaluate Kinesia One compliance in the home.

DETAILED DESCRIPTION:
In Clinic:

Participants will arrive at the clinic with deep brain stimulation (DBS) turned on and on any previously prescribed Parkinson's disease (PD) medication. Motion sensor units will be placed on the index finger, thumb, and wrist of the participant's more affected hand. The participant will then perform three repetitive motion tasks and two tremor evaluation tasks, each performed for 15 seconds. The tasks will include repetitive finger-tapping, hand opening-closing, and pronation-supination, as well as arms resting and arms extended. The sequence of five tasks will be repeated (10 task performances total) so that test-retest reliability can be examined.

The participant's DBS system will then be turned off. The two repetitions of five motor tasks will then be repeated 10 minutes, 20 minutes, and 30 minutes after DBS is turned off to measure the after-effects of DBS washout. During all task performances, motion data will be streamed from the motion sensors to a nearby computer for storage. The participant's hand will be videoed for subsequent clinical scoring. After each set of assessments (on and three time points after turning DBS off), participants will be asked to rate his/her "slowness of movement" on a 0-4 scale. The participant's DBS system will then be turned back on before he/she leaves the clinic.

To examine test-retest reliability, motion sensor-based scores will be compared to the clinician ratings. Videos from participants at both sites will be randomized, and presented to movement disorder neurologists for clinical rating. The clinician will be blinded to the participant's identity as much as possible by obscuring everything other than the participant's hand.

At Home:

Before data collection begins, a technician will give the participant a Kinesia One system (one motion sensor unit, inductive charge-pad, and tablet computer) to take home and train him/her on use. The movement tasks to be performed will be explained in detail to ensure the participant is familiar with them. The participant will be required to perform the tasks using the system twice independently before leaving the clinic to ensure he/she fully understands how to use the system. The time it takes the participant to independently set up the system will be recorded. The system will be used for two weeks, after which it will be returned to the clinic either in person or in a pre-paid shipping box.

During the two-week data collection, participants will perform a motor assessment three days per week (six days total). On each assessment day, assessments will be performed six times per day, spaced approximately two hours apart. All assessments will be performed with DBS turned ON. To begin each assessment, the participant will sit in front of the tablet computer. The software will guide the participant through the data collection procedure. The participant will be instructed to remove the motion sensor unit from the charge pad and place it appropriately on the index finger of the more affected hand. Software will then guide the participant through the assessment, which will consist of the three repetitive motion tasks and two tremor evaluation tasks, each performed for 15 seconds. The sequence of five tasks will be repeated a second time (10 task performances total) so that test-retest reliability can be examined. All data will be uploaded to a secure server. After each assessment, participants will enter rating corresponding to their perceived slowness of movement and Parkinson's state. Each week of paper diaries will be mailed back within three days after being completed in provided, pre-addressed and stamped envelopes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease
* Has Deep Brain Stimulation Implant for Parkinson's disease
* Historical bradykinesia rating of 2 or greater on at least one of the Unified Parkinson's Disease Rating Scale (UPDRS) finger-tapping, hand-movements, and pronation-supination tasks with DBS off.

Exclusion Criteria:

* Dementia (MoCA < 25)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with implanted deep brain stimulation systems for treating Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dustin A Heldman, PhD, Principal Investigator — Great Lakes NeuroTechnologies
Locations (2):
- United States (2):
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants
Started | 32
Completed | 30 (All 32 participants completed the in-clinic portion and 30 out of the 32 completed the home portion.)
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Participants
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Kinesia One Assessments Performed
Description: Percentage of Kinesia One assessments performed as directed
Time Frame: Two weeks
Measure: Mean (Standard Deviation); unit: percentage of home assessments completed
Arm/Group | Participants
Number analyzed (Participants) | 30
percentage of home assessments completed | 99 (2)

ADVERSE EVENTS:
Arm/Group | Participants
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less